CLINICAL TRIAL: NCT05865470
Title: Sex- and AGE-dependent Effects of Smoked and Oral Delta-9-THC
Brief Title: Age-dependent Effects of Smoked and Oral Delta-9-THC
Acronym: SAGE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Ziva D. Cooper, PhD, Professor / Director, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 22-001292; R01DA057252 (NIH)
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Pain; Abuse, Drug; Intoxication; Cannabinoids
Keywords: Pain; Cannabis; Delta-9-THC; Age; Sex
MeSH Terms: conditions — Pain; Substance-Related Disorders; Marijuana Abuse; Coitus | interventions — nabiximols; Dronabinol

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled study. All participants will complete all dose conditions in a randomized order.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo Comparator: Placebo (Placebo Comparator): Smoked Cannabis (0 mg THC) Oral placebo (0 mg THC)
  Interventions: Drug: Smoked Placebo; Drug: Oral Placebo
- Experimental: Low strength cannabis (Experimental): Smoked Cannabis (10 mg THC) Oral placebo (0 mg THC)
  Interventions: Drug: Cannabis; Drug: Oral Placebo
- Experimental: Higher strength cannabis (Experimental): Smoked Cannabis (20 mg THC) Oral placebo (0 mg THC)
  Interventions: Drug: Cannabis; Drug: Oral Placebo
- Experimental: Low strength oral THC (Experimental): Smoked Cannabis (0 mg THC) Oral THC (10 mg THC)
  Interventions: Drug: Dronabinol; Drug: Smoked Placebo
- Experimental: Higher strength oral THC (Experimental): Smoked Cannabis (0 mg THC) Oral THC (20 mg THC)
  Interventions: Drug: Dronabinol; Drug: Smoked Placebo

INTERVENTIONS:
Drug: Cannabis — smoked cannabis
  Other Names: Smoked cannabis with THC
  Arms: Experimental: Higher strength cannabis; Experimental: Low strength cannabis
Drug: Dronabinol — Oral delta-9-THC
  Other Names: Delta-9-THC
  Arms: Experimental: Higher strength oral THC; Experimental: Low strength oral THC
Drug: Smoked Placebo — Placebo Cannabis
  Other Names: Placebo smoked cannabis (no THC)
  Arms: Experimental: Higher strength oral THC; Experimental: Low strength oral THC; Placebo Comparator: Placebo
Drug: Oral Placebo — Oral Placebo
  Arms: Experimental: Higher strength cannabis; Experimental: Low strength cannabis; Placebo Comparator: Placebo

SUMMARY:
This study will assess the age-dependent effects of smoked and oral THC on abuse liability, intoxication, analgesia and impairment as a function of age.

DETAILED DESCRIPTION:
The overall objective of this placebo-controlled, outpatient study is to compare the dose-dependent effects of smoked and oral THC on analgesia and endpoints directly related to adverse consequences of use including abuse liability, intoxication, and impairment as a function of age and sex.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female aged 18-65 years according to the below criteria: EMERGING ADULTS: 18-25 years of age (+/- one year) MIDDLE-AGED ADULTS: 35-45 years of age (+/- one year) LATE MIDDLE-AGED ADULTS: 55-65 years of age (+/- one year)
* Report weekly-monthly use of cannabis (with primary mode of use via inhalation) over the past 6 months prior to screening
* Not currently seeking treatment for their cannabis use
* No reported clinically significant adverse effects with cannabis use
* Have a Body Mass Index from 18.5 - 34kg/m2
* Able to perform all study procedures
* FEMALES: Currently practicing an effective form of birth control if pre-menopausal

Exclusion Criteria:

* Meeting DSM-5 (Diagnostic and Statistical Manual of Mental Disorders-5) criteria for any substance use disorder other than nicotine and mild cannabis use disorder
* Report using other illicit drugs in the prior 4 weeks
* Evidence of severe psychiatric illness (e.g. mood disorder with functional impairment or suicide risk, schizophrenia) or medical condition (i.e., hypertension) judged by the study physician (and PI to put the participant at greater risk of experiencing adverse events due to completion of study procedures, interfere with their ability to participate in the study, or their capacity to provide informed consent.
* Current predominant licit use of medical cannabis
* Current use of prescription or regular use of over the counter medications (with the exception of hormonal contraceptives and hormone replacement therapy). Current use of herbal supplements that may affect study outcomes or interact with study drug (i.e., St Johns wort, kava, L-tryptophan, melatonin)
* If medical history, physical and psychiatric examination, or laboratory tests performed during the screening process are not within the normal range and / or reveal any significant illness (e.g., hypertension) as judged by the study physician and to put the participant at greater risk of experiencing adverse events due to completion of study procedures
* Current pain
* Pregnancy is exclusionary due to the possible effects of the study medication on fetal development
* History of an allergic reaction or adverse reaction to cannabis is exclusionary.
* Currently enrolled in another research protocol
* Not using a contraceptive method (hormonal or barrier methods)
* The evaluating physician reviews all medical assessments along with medical history. Any disorders that might make cannabis administration hazardous are exclusionary.
* Intolerance to lactose and sesame (ingredients in the oral THC preparation)
* Insensitivity to the Cold Pressor Test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2028-10-15 (Estimated); Study Completion 2029-10-15 (Estimated)

PRIMARY OUTCOMES:
Subject-rated drug effects | 6 hours
  Average and peak subjective ratings of drug effects associated with abuse liability and intoxication as measured using visual analogue scales (VAS; 1-100mm).
Analgesia as measured using the Cold Pressor Test | 6 hours
  Peak and average pain threshold and tolerance assessed using the Cold Pressor Test
Impairment | 6 hours
  The primary outcome measure for performance will be the peak difference from baseline scores of the Global Impairment Score
Pharmacokinetics of THC and metabolites | 6 hours
  Plasma levels of THC, 11-OH-THC, and THCCOOH

CONTACTS AND LOCATIONS:
Overall Officials: Ziva Cooper, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Cannabis and Cannabinoids, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No